CLINICAL TRIAL: NCT06727643
Title: Comparison of Acute Effects of Flexible and Rigid Taping on Core Strength in Healthy Young Adults: A Randomized Controlled Trial
Brief Title: Comparison of Acute Effects of Flexible and Rigid Taping on Core Strength in Healthy Young Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Esra BAYRAMOĞLU DEMİRDÖĞEN, lecturer, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KAEU-EBAYRAMOGLUD-002
Record Dates: First submitted 2024-11-10; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Trunk Muscle Strength
Keywords: core muscle strength; elastic tape; rigid tape

STUDY DESIGN:
Intervention Model Description: 2 different tape types will be applied to 2 different groups and the results will be compared.
Who Masked: Outcomes Assessor
Masking Description: The researcher taking the measurements will not be aware of the application made.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- elastic tape group (Other): Participants in this group will have their core muscles taped with flexible tape.
  Interventions: Other: trunk muscle strength; Other: Core Strength; Other: Balance
- rigid tape group (Active Comparator): Participants in this group will have their core muscles taped with rigid tape.
  Interventions: Other: trunk muscle strength; Other: Core Strength; Other: Balance

INTERVENTIONS:
Other: trunk muscle strength — force that represents the endurance of the body.
Other: Core Strength — back and abdominal muscle endurance
Other: Balance — steady state

SUMMARY:
Trunk stabilization refers to the optimization of posture for conscious and unconscious movements, the maintenance of upright posture, and the stabilization of arm and head movements.

Trunk stabilizer muscles reduce overload between the intervertebral joints and play an important role in maintaining the stability of the spine. Trunk stabilizer muscles are connected via fascia, and superficial and deep muscles control the positions of the trunk to facilitate trunk stabilization.

Prolonged activity of trunk stabilization muscles causes fatigue in one or more muscles, which can lead to loss of neuromuscular control and cause tissue damage and back pain due to uncontrolled movements.

Muscular fatigue is defined as a decrease in the maximum strength or strength capacity of muscles after continuous physical activity. Sore or weak muscles tend to fatigue more quickly, which leads to a decrease in the ability to perform physical activities. When the endurance of the trunk stabilizer muscles decreases due to muscle fatigue, concentric and eccentric signal patterns are disrupted, causing the muscles to react less quickly. Muscle fatigue also reduces exercise performance and increases the risk of pain and injury. Therefore, increasing muscle endurance in cases of spinal instability may be more important than muscle strength training. Recently, flexible tape has begun to be used in the treatment of muscle fatigue. Taping has been used for years in both athletes and physiotherapy clinics for reducing pain, preventing injuries, biomechanical correction, increasing stability, increasing proprioception, reducing edema, as well as muscle inhibition and facilitation. Recently, taping techniques that primarily aim to change muscle activity have become widespread physiotherapy methods. In particular, it has been shown that taping inhibits or facilitates the muscle by changing the muscle's reflex amplitude (H reflex). When the literature is examined, it is seen that studies on taping are focused especially on flexible taping applications, and that studies on rigid taping applications are few. Therefore, in this study, the researchers aimed to compare the effects of flexible and rigid taping on trunk muscle endurance (core) and trunk stability when all trunk stabilizer muscles are used.

DETAILED DESCRIPTION:
The study will include 56 healthy individuals from the relatives of patients who are between the ages of 18-25, who have no medical history of spinal musculoskeletal disorders in the last 6 months, who do not have a current neurological or orthopedic contracture, who do not have a history of contact dermatitis or a history of cutaneous adverse reactions to flexible or rigid tape, and who have not been diagnosed with scoliosis or a herniated disc in the last 6 months and who agree to participate in the study.

The trunk muscle strength (core) of all individuals participating in the study will be evaluated with the McGill Core Endurance Tests and the Sharman Test, and their stability-balance with the Biodex Balance System (does not contain radiation or similar harmful rays) with eyes open and closed.

The individuals will be divided into two groups using the envelope drawing method and will be subjected to trunk endurance tests and trunk stability tests before taping. Flexible taping will be applied to one group and rigid taping will be applied to the other, and endurance tests and stability tests will be repeated immediately after taping. Tapings and measurements will be performed by different physiotherapists to ensure blindness.

The tapes investigators will use are the ones that people apply themselves, even on internet sites, and do not harm the person or the environment. The tapes will be applied by a specialist physiotherapist, will remain on the patient for the duration of the evaluations (20 minutes on average) and will be removed by the physiotherapist when the evaluations are over. The tapes will not be left on the participant.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25,
* not having a medical history of musculoskeletal disorders of the spine in the last 6 months,
* not having a current neurological or orthopedic contracture,
* not having a history of contact dermatitis or cutaneous adverse reactions to flexible or rigid tape,
* not having been diagnosed with scoliosis or a herniated disc in the last 6 months,
* being willing to participate in the study

Exclusion Criteria:

* Not being between the ages of 18-25,
* having a medical history of musculoskeletal disorders of the spine within the last 6 months,
* having current neurological or orthopedic contracture,
* having a history of contact dermatitis or a history of cutaneous adverse reactions to flexible and rigid tape,
* having been diagnosed with scoliosis or a herniated disc within the last 6 months,
* not volunteering to participate in the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Trunk Muscle Strength | 15 minutes before taping and 15 minutes after taping
  Trunk Flexion Test: The participant is asked to cross their hands over their chest. They are positioned on the floor with their trunk at 60° flexion and their knees at 90° flexion. The time until there is any deterioration in their position is recorded. The same test is applied for trunk extension and right-left bridge positions and the times are recorded.
Core Strength | 20 minutes before taping and 20 minutes after taping
  Sharman Test: The participant is lying in the supine position and the stabilizer is placed on the natural lordotic curve, the stabilizer pressure is adjusted to 40 mmHg by the physiotherapist performing the test, and then the abdominal bracing maneuver is taught to the participant. This maneuver provides isolated contraction of the transversus abdominus muscle and spinal stability. The test consists of 5 stages. The person being tested is asked to perform the abdominal bracing maneuver at each stage of the test and to perform different lower extremity movements while continuing this maneuver. The difficulty level of the test increases from level 1 to level 5. A value change of more than 10 mmHg in the stabilizer during each stage movement means that the patient has not completed that level and the test is terminated.

SECONDARY OUTCOMES:
balance | 10 minutes before taping and 10 minutes after taping
  Stability - Balance: The patient will be positioned on a platform with a screen in front of them. In our study, a rigid platform will be used and the patient will be given a suitable position by holding on to the side bars with their hands while both feet (bare) are on the platform. The foot coordinates are determined while the patient is in the most comfortable position where they can maintain their balance. For static postural balance measurement, patients are asked to hold the circular ring they see on the screen in the center for 20 seconds. The test is terminated after 3 measurements including 10-second rest periods. Patients will repeat this measurement with their eyes open and closed.

CONTACTS AND LOCATIONS:
Overall Officials: AHİ EVRAN UNIVERSITY, Study Chair — KIRŞEHİR AHİ EVRAN PHYSICAL THERAPY AND REHABILITATION HOSPITAL
Locations (1):
- Kirşehir Ahi Evran University Physical Therapy and Rehabilitation Hospital, Kırşehir, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No